CLINICAL TRIAL: NCT05203536
Title: ICEBERG STUDY. Respiratory Mechanics Assessment During Assisted Mechanical Ventilation
Brief Title: Respiratory Mechanics Assessment During Assisted Mechanical Ventilation
Acronym: ICEBERG
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: 3552
Record Dates: First submitted 2021-12-23; First posted 2022-01-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Hypoxemic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To verify the association between respiratory system mechanical properties (ΔP, ΔPL,dyn, Pmus, Pplat and CRS and CL,dyn) assessed during assisted modes of ventilation (as average over the first three days since enrollment) and ICU mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute Hypoxaemic Respiratory Failure (defined as respiratory failure requiring invasive mechanical ventilation with a PaO2/FiO2< 300 mmHg) during the course of ICU stay (including ARDS).
* Invasive mechanical ventilation in one of these modes: Pressure A/C, PRVC, SIMV PC, PSV, NAVA, PAV+, BiPAP
* Presence of spontaneous breathing activity (ventilator triggering), since 6 hours and no longer than 48 hours
* Patient for full active management at this point.

Exclusion Criteria:

* Age <18 years old
* Pregnancy
* Active air leaks
* Moribund state
* High ICP
* Patient has passed a spontaneous breathing trial (if performed for clinical indication)
* Known COPD with history of home oxygen therapy and/or non invasive ventilation and/or GOLD III-IV. Non invasive ventilation for sleep apnea is NOT an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AHRF/ARDS patients on Assisted Mechanical Ventilation modes from international centers will be enrolled. All the pressure-targeted modes of assisted ventilation will be acceptable for the study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Correlation between respiratory system mechanical properties and ICU mortality | 90 days
  Difference between mean values of driving pressure in survivors and non-survivors at ICU discharge.

SECONDARY OUTCOMES:
Correlation between respiratory system compliance and ICU mortality | 90 days
  Difference between mean values of respiratory system compliance in survivors and non-survivors at ICU discharge.
Correlation between plateau pressure and ICU mortality | 90 days
  Difference between mean values of plateau pressure in survivors and non-survivors at ICU discharge.
Correlation between pressure muscle index and ICU mortality | 90 days
  Difference between mean values of pressure muscle index (PMI) in survivors and non-survivors at ICU discharge.
Correlation between muscle pressure and ICU mortality | 90 days
  Difference between mean values of muscle pressure (Pmus) in survivors and non-survivors at ICU discharge.

CONTACTS AND LOCATIONS:
Locations (8):
- Toronto General Hospital, Toronto, Toronto, Canada
- University Medical Centre Schleswig-Holstein, Kiel, Kiel, Germany
- University Hospital Galway, Galway, Galway, Ireland
- Italy (3):
  - Ospedale Sant'Anna, Ferrara, Ferrara
  - Policlinico di Milano Ospedale Maggiore, Milan, Milano
  - ASST-Monza, Ospedale San Gerardo, Monza, Monza
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona